CLINICAL TRIAL: NCT05214664
Title: Efficacy of a Guiding Device for Inferior Alveolar Nerve Block, EZ-Block®, Compared With a Conventional "Freehand" Administration, in Providing Anesthesia During Surgical Removal of Impacted Lower Third Molar.
Brief Title: Efficiency of a Guiding Device for Inferior Alveolar Nerve Block, EZ-Block®, Compared to a Conventional Freehand Administration.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: EZ-BLOCK; 2020-A02755-34 (Other: ANSM)
Record Dates: First submitted 2022-01-17; First posted 2022-01-31 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Tooth Avulsion
MeSH Terms: conditions — Tooth Avulsion | interventions — Anesthesia

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, single-blind, controlled clinical trial with cross-over.
Who Masked: Investigator
Masking Description: In each center, a pair of practitioners has been identified: one practitioner, "Anesthesia", will be in charge of the randomization and the realization of the anesthesia by one of the two techniques (EZ-Block or conventional freehand technique). Another practitioner, "Surgery", will be blinded to the anesthesia technique used. It is this practitioner who will perform the surgical procedure described below.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guiding device for inferior alveolar nerve block (Experimental): The system consists of a reusable angulator with a tube, a reusable plunger, and a single-use syringe body.
  These three components are combined with a single-use needle and an anesthetic cartridge to create the ready-to-use EZ-Block® device.
  Interventions: Procedure: Anesthesia
- Conventional freehand technique for providing anesthesia (Active Comparator): The injection site is located in the middle of the triangle with an upper base formed, during maximum mouth opening, outside by the mandibular ramus, inside by the mesial pterygoid muscle and above by the lateral pterygoid muscle.
  The needle is inserted up to the bone contact (about 20mm) while the body of the syringe is directed towards the contralateral premolars or molars.
  Use of a disposable carpule syringe with aspiration. Use of a 35mm long needle with a 0.5mm diameter. Use of an articaine anesthesia carpule with adrenaline 1/200000.
  Interventions: Procedure: Anesthesia

INTERVENTIONS:
Procedure: Anesthesia — Once the anesthesia is performed by the "Anesthesia" practitioner either with the EZ-Block® device or by the conventional freehand technique, the surgical procedure will be performed in the same way in both arms, and for each tooth, by the "Surgery" practitioner:
  * The "Surgery" practitioner takes charge of the patient after a post-anesthesia time of 10 minutes and performs a new antisepsis then completes the anesthesia by anesthetizing the buccal and lingual nerve with a carpule of 1.8ml of articaine + adrenaline at 1/200000.
  * The "Surgery" practitioner starts the surgical procedure.
  * In the absence of pain, the practitioner "Surgery" carries out the surgical act in its totality (situation of success for the principal criterion of the study) then records the EVA at the end of the intervention.

SUMMARY:
The success rates reported in the literature for the various truncal anesthesia techniques are extremely variable and have shown a lack of reproducibility of the techniques. The use of the EZ-BLOCK® guidance system would increase this success rate in a significant and reproducible way, as it is based on individualized anatomical foundations and therefore adapted to inter-patient variability.

In order to determine its effectiveness in clinical situations encountered in current practice, a comparative clinical study of the 2 techniques (freehand reference technique and using the EZ-BLOCK® system) is necessary.

DETAILED DESCRIPTION:
The use of loco-regional anesthesia in the mandibular foramen (Inferior Alveolar Nerve Block - IANB) is part of the therapeutic arsenal for any Dental Surgeon or specialist in Oral Surgery or Endodontics. These local-regional anesthesias are indicated for restorative, endodontic and single and/or multiple surgical treatments of mandibular teeth homolateral to the infiltrated side. The so-called "conventional" freehand reference technique was described by William Steward Halsted and compared in numerous studies to other truncal anesthesia techniques such as Gow Gates or even Akinosi-Vazirani.

Certain anatomical landmarks must be accurately identified by the operator to reduce the percentage of failure of this technique. Conventional IANB is associated with a 40% failure rate in surgical removal of the lower third molars included, which is the highest percentage of all clinical failures obtained under local anesthesia.

The purpose of this study is to compare the success rate of a IANB guidance device, EZ-Block®, with traditional freehand anatomic administration in the surgical removal of impacted lower third molars.

The use of the EZ-BLOCK® guidance system would increase the success rate significantly and reproducibly because it is based on individualized anatomical foundations and is therefore adapted to inter-patient variability.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years of age or older
2. Dental panoramic radiograph or cone beam examination less than 6 months prior to inclusion
3. Clinical criteria and similar radiographs of the 2 mandibular third molars:

   1. Stage of root planing
   2. Normoposition, horizontal
   3. Type of eruption: disincluded, impacted, impacted
   4. Anatomical relationship between inferior alveolar nerve and mandibular wisdom tooth apices similar for both sides
4. Affiliation to a social security scheme
5. Informed consent, dated and signed before any study procedure is performed

Exclusion Criteria:

1. Pregnant or breastfeeding woman
2. Known allergy to the anesthetic molecule or to a component of the anesthetic carpule
3. Contraindication to the use of vasoconstrictor in dental anesthesia
4. Contraindication to a therapeutic procedure under local anesthesia
5. Patients taking TKA for another medical reason
6. Presence of a cystic pathology related to at least 1 of the 2 mandibular third molars to be extracted
7. Limitation of mouth opening
8. Associated systemic pathology requiring priority management
9. Inability of the patient to comply with study follow-up and scheduled visits (especially for second wisdom tooth avulsion)
10. Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The success of the truncal infiltration of anesthetic product will be defined as the absence of recourse to additional anesthesia during the procedure | During the procedure
  The success of the truncal infiltration of anesthetic product will be defined as the absence of recourse to additional anesthesia during the procedure (binary criterion yes / no).

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) of pain | During the procedure
  Visual Analog Scale (VAS) of pain
Total cumulative dose of anesthetic used | During the procedure
  Total cumulative dose of anesthetic used
Adverse event report | Up to 10 days after the second intervention
  adverse event report

OTHER OUTCOMES:
The success of the truncal infiltration of anesthetic product will be compared by center | During the procedure
  The success rate of the truncal infiltration of anesthetic product will be compared by center

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Alix Fauroux, MD, Study Director — CHU Montpellier - UFR Odontologie de Montpellier
Locations (5):
- France (5):
  - CHU Montpellier, Montpellier
  - CHRU Nancy Service d'odontologie Brabois adultes, Nancy
  - Service de médecine bucco-dentaire Hôpital BRetonneau - APHP, Paris
  - Hôpitaux universitaires de Strasbourg Hôpital Civil Pôle de Médecine et chirurgie bucco-dentaires, Strasbourg
  - Odontologie et traitement dentaire Pôle clinique des voies respiratoires Faculté de chirurgie dentaire, Toulouse

REFERENCES:
- [Background] Haas DA. Alternative mandibular nerve block techniques: a review of the Gow-Gates and Akinosi-Vazirani closed-mouth mandibular nerve block techniques. J Am Dent Assoc. 2011 Sep;142 Suppl 3:8S-12S. doi: 10.14219/jada.archive.2011.0341. PMID 21881056
- [Background] Ravi Kiran BS, Kashyap VM, Uppada UK, Tiwari P, Mishra A, Sachdeva A. Comparison of Efficacy of Halstead, Vazirani Akinosi and Gow Gates Techniques for Mandibular Anesthesia. J Maxillofac Oral Surg. 2018 Dec;17(4):570-575. doi: 10.1007/s12663-018-1092-5. Epub 2018 Feb 26. PMID 30344402
- See also: Alternative mandibular nerve block techniques: a review of the Gow-Gates and Akinosi-Vazirani closed-mouth mandibular nerve block techniques — https://pubmed.ncbi.nlm.nih.gov/21881056/
- See also: Comparison of Efficacy of Halstead, Vazirani Akinosi and Gow Gates Techniques for Mandibular Anesthesia — https://pubmed.ncbi.nlm.nih.gov/30344402/